CLINICAL TRIAL: NCT04169620
Title: Effectiveness of a Program With Aquatic Therapy in Patients With Parkinson's Disease Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, SAGRARIO PÉREZ DE LA CRUZ, Clinical Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: spd205
Record Dates: First submitted 2016-11-02; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease; Physical Disability
MeSH Terms: conditions — Parkinson Disease | interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- variable aquatic Ai Chi (Experimental): The 15 patients assigned to the aquatic therapy group (experimental group) received 20 twice-weekly sessions in total, during the same period of time as the control group. These 20 sessions consisted of group sessions lasting 45-minutes.
  The sessions were designed with a gradual increase in difficulty. Initially, a recreational warm-up activity was performed, followed by 30 minutes dedicated to practicing the Ai Chi Program. At the end of the session there was a calming down activity. The exercises were performed in a specific order, until completion of the 19 possible movements.
  Interventions: Other: aquatic Ai Chi
- variable dry land (Placebo Comparator): These sessions consisted of group sessions of supervised training lasting 45 minutes each. These comprised a 10-minute warm-up that included exercises for gait, trunk mobility and exercises involving the upper and lower limbs. The central part of the sessions consisted of 30-40 minutes of strength training and aerobic exercises, both individual and in groups. Each session was performed with a specific intensity goal, in order to end with a cooling down period, comprising 20 minutes of functional exercises based on activities of daily living, balance exercises, facial muscle exercises, proprioceptive exercises, muscle relaxation and stretching.
  Interventions: Other: control

INTERVENTIONS:
Other: aquatic Ai Chi — The sessions took place in a pool measuring 20 m x 6 m, at a depth of 110 cm. The water temperature was 30oC (with variations of less than 0.5o) and the room temperature was 27.5oC (with variations of less than 1o). The proportions of the pool were ideally suited for collective treatment.
  The sessions were designed with a gradual increase in difficulty. Initially, a recreational warm-up activity was performed, followed by 30 minutes dedicated to practicing the Ai Chi Program. At the end of the session there was a calming down activity. The exercises were performed in a specific order, until completion of the 19 possible movements.
  Arms: variable aquatic Ai Chi
Other: control — These sessions consisted of group sessions of supervised training lasting 45 minutes each. These comprised a 10-minute warm-up that included exercises for gait, trunk mobility and exercises involving the upper and lower limbs. The central part of the sessions consisted of 30-40 minutes of strength training and aerobic exercises, both individual and in groups. Each session was performed with a specific intensity goal, in order to end with a cooling down period, comprising 20 minutes of functional exercises based on activities of daily living, balance exercises, facial muscle exercises, proprioceptive exercises, muscle relaxation and stretching.
  Arms: variable dry land

SUMMARY:
The aim of this study is to determine the effect of an aquatic Ai Chi training program on the perception of pain, the maintenance of balance and the functional independence of patients with Parkinson's disease.

Fifteen patients diagnosed with Parkinson's disease (Hoehn and Yahr range: 1-3) participated in a program of Aquatic Ai Chi lasting ten weeks with sessions held twice weekly. These were compared to a group of 15 Parkinson patients (control group) who received therapy on dry land.

DETAILED DESCRIPTION:
All study participants met the following inclusion criteria: individuals diagnosed with PD in stages 1 to 3 (Hoehn and Yahr Scale), older than 40 years, in the off phase (not medicated) and with a score greater or equal to 24 on the Mini-Mental State Examination Scale, without any medical contraindications and who accepted the study norms (regular assistance and active participation). The exclusion criteria were: individuals who did not comply with the above mentioned criteria, and the presence of articular and/or muscular lesions in the lower limbs affecting independent gait.

The procedure of randomization was performed for the overall sample using stratified randomization controlling for the Hoehn & Yahr stage employing Excell software (Microsoft Excell 2013: Microsoft Corp. Redmond WA).

The participants received an initial assessment on dry land lasting 30-45 minutes, performed by a physiotherapist not involved in the study. Timetable norms were disclosed as well as recommendations regarding appropriate clothing for the activity. A baseline assessment was performed prior to commencing therapy. This was repeated upon completion of all sessions while a follow-up assessment took place one month later.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with PD in stages 1 to 3 (Hoehn and Yahr Scale), older than 40 years, in the off phase (not medicated) and with a score greater or equal to 24 on the Mini-Mental State Examination Scale, without any medical contraindications and who accepted the study norms (regular assistance and active participation).

Exclusion Criteria:

* individuals who did not comply with the above mentioned criteria, and the presence of articular and/or muscular lesions in the lower limbs affecting independent gait.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain assessed with VAS scale | ten weeks
  VAS scale

SECONDARY OUTCOMES:
Balance assessed with Berg Balance scale | ten weeks
  Berg Balance scale
Functionality assessed with UPDRS scale | ten weeks
  UPDRS scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Almería, La Cañada de San Urbano, Almería, Spain

IPD SHARING:
Plan to Share IPD: Undecided